CLINICAL TRIAL: NCT01698749
Title: Effect of Intravitreal Long Acting Dexamethasone Implant, Ozurdex in Patients With Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Pooja Bansal,MD, MD, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PoojaBansal 13
Record Dates: First submitted 2012-03-22; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Macular Edema; Macular Edema, Cystoid; Vision Disorders; Clinically Significant Macular Edema
Keywords: Ozurdex; Diabetic macular edema; Central macular thickness
MeSH Terms: conditions — Macular Edema; Vision Disorders | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ozurdex in diabetic macular edema (Experimental): Intravitreal ozurdex given in patients with diabetic macular edema and patients followed up for change in central macular thickness and visual acuity over period of 6 months
  Interventions: Drug: long acting intravitreal dexamethasone implant

INTERVENTIONS:
Drug: long acting intravitreal dexamethasone implant — Intravitreal ozurdex was given in diabetic patients with clinically significant macular edema and they were followed up for change in central macular thickness and visual acuity over a period of 6 months
  Other Names: Ozurdex

SUMMARY:
This study is undertaken to determine the effect of intravitreal long acting dexamethasone implant,(Ozurdex®)in patients with diabetic macular edema.Diabetic macular edema is important cause of visual impairment in patients with diabetes mellitus. Focal/ grid laser photocoagulation is the standard of care in its management. Several adjuncts including intravitreal corticosteroids, Pegabtanib Sodium ,Ranibizumab, Bevacizumab, non-steroidal anti-inflammatory agents, corticosteroids, laser photocoagulation have been tried. Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern as the patients need multiple repeat injections because of its short half life. A more potent steroid, dexamethasone has also been tried as an alternative to TA for macular edema; however, its short half life of only 3 hours prevents its clinical application. In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (Dexamethasone DDS - Ozurdex®, Allergan Inc, Irvine, California) was recently developed. Promising results have been shown in certain patients with retinal vein occlusions, uveitis receiving this intravitreal drug delivery system with improvement in visual acuity. The present study introduces a novel concept of using Ozurdex ® implant in patients with diabetic macular edema.

DETAILED DESCRIPTION:
This study is undertaken to determine the effect of intravitreal long acting dexamethasone implant,(Ozurdex®)in patients with diabetic macular edema.Diabetic macular edema is important cause of visual impairment in patients with diabetes mellitus. Focal/ grid laser photocoagulation is the standard of care in its management. Several adjuncts including intravitreal corticosteroids, Pegabtanib Sodium ,Ranibizumab, Bevacizumab, non-steroidal anti-inflammatory agents, corticosteroids, laser photocoagulation have been tried. Intravitreal Triamcinolone Acetonide (TA), a water insoluble steroid, has been shown to reduce the retinal thickness and improve the visual acuity. However, recurrence of macular edema in patients who receive intravitreal TA is a major concern as the patients need multiple repeat injections because of its short half life. A more potent steroid, dexamethasone has also been tried as an alternative to TA for macular edema; however, its short half life of only 3 hours prevents its clinical application. In search for the ideal corticosteroid preparation, a Dexamethasone Posterior Segment Drug Delivery System (Dexamethasone DDS - Ozurdex®, Allergan Inc, Irvine, California) was recently developed. Promising results have been shown in certain patients with retinal vein occlusions, uveitis receiving this intravitreal drug delivery system with improvement in visual acuity. The present study introduces a novel concept of using Ozurdex ® implant in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* The patients of Type 1 or Type 2 Diabetes Mellitus fulfilling the following inclusion criteria shall be enrolled in the study:

  1. Patients of Non Proliferative Diabetic retinopathy (NPDR)with clinicaly significant macular edema(CSME)
  2. Patients with Proliferative Diabetic Retinopathy (PDR) with CSME where proliferative component has been adequately treated with laser photocoagulation
  3. Diabetic patients withcystoid macular edema
  4. Minimum central thickness on OCT not less than 300 microns

Exclusion Criteria:

1. Patients with history of ocular hypertension or glaucoma
2. Patients with media haze or pupillary non-dilation that does not allow good fundus photography, FFA and OCT.
3. Patients with macular ischemia on FFA

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change in central macular thickness | Baseline and 6 months
  The primary outcome is the change in the central macular thickness, either an increase or decrease, as measured by optical coherence tomography as compared to baseline central macular thickness

SECONDARY OUTCOMES:
Change in the visual acuity | Baseline and 6 months
  Change in the visual acuity as measured by the logMAR visual acuity chart

CONTACTS AND LOCATIONS:
Overall Officials: POOJA BANSAL, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; VISHALI R GUPTA, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; AMOD GUPTA, MBBS,MS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Pooja Bansal, Chandigarh, Chandigarh, India